CLINICAL TRIAL: NCT05565885
Title: Search for BIO Diagnostic and Prognostic Markers in Adult VAScularitis
Acronym: BIOVAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220193-BIOVAS
Record Dates: First submitted 2022-09-07; First posted 2022-10-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Vasculitis
Keywords: biomarkers; diagnosis; prognosis
MeSH Terms: conditions — Vasculitis; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sampling at diagnosis, at M1, M3, M12 and at the time of a possible relapse: 14 ml of additional blood during a blood puncture for routine care will be collected at each visit together with clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with vascularitis: Two additional 7ml EDTA tubes of blood are taken from the same blood puncture as during routine follow-up at several points in the follow-up
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — 4 blood sampling per patient and an additional one in case of relapse

SUMMARY:
To date, there are no reliable diagnostic blood markers of adult vasculitis. To date, the diagnosis of vasculitis is based on invasive procedure, biopsy of affected tissues potentially at risk of complication . In addition, there are no reliable biomarkers to predict the evolution of vasculitis (relapse, refractory form ...) necessary for the management of patients (type of treatment, duration ..)

Prospective study, monocentric (CHU de Tours), non-interventional, aimed at finding diagnostic and prognostic biomarkers (both metabolomic and immunologic) in adult vasculitis patients.

DETAILED DESCRIPTION:
Specimen will be collected at diagnosis, month 1, month 3, and month12 and at the time of a possible relapse. 14 ml of additional blood during a blood puncture made for routine care will be collected at each visit as well as clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Active vasculitis, new diagnosis or relapse
* IgA vasculitis
* ANCA vasculitis
* Giant cell arteritis

Exclusion Criteria:

* Person who has objected to the processing of data
* Pregnant woman
* Patient positive for HIV, HBV, HCV
* Treatment in the previous month with corticosteroids, immunosuppressive drugs or biotherapy.
* Patient unable to understand the information leaflet
* Adult under guardianship or curatorship

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with vascularitis
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2037-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
cytokine/chemokine/metabolite concentrations | Baseline
  Analysis by méthod Luminex
cytokine/chemokine/metabolite concentrations | Month 1
  Analysis by méthod Luminex
cytokine/chemokine/metabolite concentrations | Month 3
  Analysis by méthod Luminex
cytokine/chemokine/metabolite concentrations | Month 12
  Analysis by méthod Luminex
cytokine/chemokine/metabolite concentrations | date of relapse assessed up to 12 months
  Analysis by méthod Luminex
percentage of different non-conventional T cell populations | Baseline
  study by flow cytometry
percentage of different non-conventional T cell populations | Month 1
  study by flow cytometry
percentage of different non-conventional T cell populations | Month 3
  study by flow cytometry
percentage of different non-conventional T cell populations | Month 12
  study by flow cytometry
percentage of different non-conventional T cell populations | date of relapse assessed up to 12 months
  study by flow cytometry

SECONDARY OUTCOMES:
cytokine/chemokine/metabolite concentrations | baseline
  identify a metabolomic blood profile for the prognosis of vasculitis
cytokine/chemokine/metabolite concentrations | Month 1
  identify a metabolomic blood profile for the prognosis of vasculitis
cytokine/chemokine/metabolite concentrations | Month 3
  identify a metabolomic blood profile for the prognosis of vasculitis
cytokine/chemokine/metabolite concentrations | Month 12
  identify a metabolomic blood profile for the prognosis of vasculitis
cytokine/chemokine/metabolite concentrations | date of relapse assessed up to 12 months
  identify a metabolomic blood profile for the prognosis of vasculitis
percentage of different non-conventional T cell populations | baseline
  identify an immunological blood profile for the prognosis of vasculitis
percentage of different non-conventional T cell populations | Month 1
  identify an immunological blood profile for the prognosis of vasculitis
percentage of different non-conventional T cell populations | Month 3
  identify an immunological blood profile for the prognosis of vasculitis
percentage of different non-conventional T cell populations | Month 12
  identify an immunological blood profile for the prognosis of vasculitis
percentage of different non-conventional T cell populations | date of relapse assessed up to 12 months
  identify an immunological blood profile for the prognosis of vasculitis
metabolomic pathway | baseline
  Identify a metabolomic pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
metabolomic pathway | Month 1
  Identify a metabolomic pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
metabolomic pathway | Month 3
  Identify a metabolomic pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
metabolomic pathway | Month 12
  Identify a metabolomic pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
metabolomic pathway | date of relapse assessed up to 12 months
  Identify a metabolomic pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
immunological pathway | baseline
  Identify an immunological pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
immunological pathway | Month 1
  Identify an immunological pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
immunological pathway | Month 3
  Identify an immunological pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
immunological pathway | Month 12
  Identify an immunological pathway involved in the pathophysiology of vasculitis that could be a target for therapy.
immunological pathway | date of relapse assessed up to 12 months
  Identify an immunological pathway involved in the pathophysiology of vasculitis that could be a target for therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided